CLINICAL TRIAL: NCT00921635
Title: A Phase III Study to Evaluate the Impact of Maintaining Haemoglobin Levels Above 120g/L Verses Above 100g/L in Anaemic Patients With Carcinoma of the Cervix Receiving Concurrent Cisplatin and Radiation Therapy
Brief Title: A Study to Evaluate the Impact of Maintaining Hemoglobin Levels in Anemic Patients With Carcinoma of the Cervix
Acronym: HOSTT
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Yee-Min Jen/Head of the department of Radiation oncology, Radiation oncology of Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANZGOG0401; TSGHIRB095-05-044
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2009-06

CONDITIONS: Cervical Cancer; Anemia
Keywords: Haemoglobin
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anemia | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maintain hemoglobin level above 120 g/L (Experimental): Hemoglobin level from 120 g/L to 130 g/L
  Interventions: Procedure: Blood transfusion
- Maintain hemoglobin level above 100 g/L (Active Comparator): Hemoglobin level from 100 g/L to 110 g/L
  Interventions: Procedure: Blood transfusion

INTERVENTIONS:
Procedure: Blood transfusion — Blood transfusion to maintain hemoglobin level above 120 g/L
  Arms: Maintain hemoglobin level above 120 g/L
Procedure: Blood transfusion — Blood transfusion to maintain hemoglobin level above 100 g/L
  Arms: Maintain hemoglobin level above 100 g/L

SUMMARY:
The purpose of this study is to assess the feasibility, safety and short term effects on health related quality of life, of maintaining hemoglobin from 120 to 130 g/L versus from 100 to 110 g/L, with red cell concentrate (RCC) transfusion, in women having chemo-radiation for cancer of the cervix.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated cervix cancer
* FIGO stage IB2, II, IIIB, IVA
* Suitable for treatment with radical intent using concurrent cisplatin and pelvic radiation

Exclusion Criteria:

* Hemoglobin level above 125g/L
* Lower one-third vaginal involvement
* Para-aortic lymphadenopathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
The impact of maintaining hemoglobin levels above 120 g/L versus above 100 g/L | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yee-Min Jen, Principal Investigator — Randiation Oncology